CLINICAL TRIAL: NCT05615909
Title: PRO-MR-RT Systematic Web-based Patient-reported Outcomes for a Personalized, Patient-centered Symptom Management and Clinical Assessment of Pelvic Toxicity to Magnetic Resonance Radiation Therapy
Brief Title: PRO-MR-RT Systematic Patient-reported Outcomes to Pelvic Online MRgRT
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry); AgeCare Academy of Geriatric Cancer Research (Unknown)
Responsible Party: Principal Investigator, Pia Krause Møller, BN, MPH, Phd Student, Odense University Hospital
Other Study IDs: OP_775
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Acute toxicity; Patient-reported outcome
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Online MR-guided radiotherapy: Prostate cancer patients treated with online MR-guided radiotherapy in the Unity MR-linac.
  Interventions: Radiation: Online MR-guided radiotherapy
- CT-guided radiotherapy: Prostate cancer patients treated with CT-guided radiotherapy (VMAT) in linear accerelators.
  Interventions: Radiation: CT-guided radiotherapy

INTERVENTIONS:
Radiation: Online MR-guided radiotherapy — Online adaptive MR-guided radiotherapy in the Unity MR-linac for localized intermediate risk prostate cancer (60 Gy/20 fx) or low-volume metastatic prostate cancer (36 Gy/6 fx).
  Groups: Online MR-guided radiotherapy
Radiation: CT-guided radiotherapy — CT-guided radiotherapy in linear accelerators for patients with high-risk prostate cancer (78 Gy/39 fx), intermediate risk prostata cancer (60 Gy/20 Fx) or having salvage radiotherapy (70 Gy/35 fx)
  Groups: CT-guided radiotherapy

SUMMARY:
In 2018 the Unity MR-linac was approved for treating patients with online magnetic resonance (MR)-guided radiotherapy. With the MR-linac it is possible to get real-time MR images with high soft tissue contrast, adapt the radiotherapy plan and subsequently irradiate at each treatment fraction. Patients with prostate cancer is one of the patient groups referred for this new treatment and potentially they will benefit with decreased margins around the tumour and increased local tumor control rates.

The acute toxicity is important when evaluating treatment tolerability. A prospective longitudinal observation of the acute treatment toxicity to online MR-guided radiotherapy is therefore essential in the evaluation of this new technology.

Patient-reported outcomes (PRO) are disease symptoms and treatment toxicity reported directly by patients themselves without clinician interpretation. Several studies have indicated that clinicians tend to underreport the incidence and severity of patient symptoms, thus a systematic use of PROs in clinical trials can provide valuable evidence to the clinicians. As online MR-guided radiotherapy (MRgRT) is a new technology there is limited research worldwide on patient-reported symptoms and quality of life.

The objective of this study is therefore to prospectively investigate the patient-reported acute toxicity and changes in quality of life during and after online MR-guided radiotherapy.

DETAILED DESCRIPTION:
Background:

In 2018 the first patients worldwide were treated with the first 1.5 T MR-linac. The MR-linac is innovative technology in cancer treatment making precision radiotherapy possible, as it is a linear accelerator mounted on a ring around a 1.5-Tesla MRI Scanner combined with an online adaptive radiotherapy planning system. When the patient is positioned in the MR-linac it is possible to get real-time MR images with high soft tissue contrast, adapt the radiotherapy plan and subsequently irradiate at each treatment fraction. The improved visualization on the MR images makes it possible to see how the tumour and the organs around it changes and adapt the treatment plan every day. This opens up for a reduction of safety margins needed to insure target coverage and increased use of hypo- fractionation. Cancer patients will hopefully benefit from this with decreased treatment toxicity and increased local tumor control rates.

Today, computed tomography (CT)-guided intensity-modulated radiotherapy is standard treatment for patients with pelvic or abdominal tumors. However, the visualization of the tumor and surrounding tissue is poor due to low soft-tissue contrast in the cone-beam scans. When using MRI for online radiotherapy planning in pelvic and abdominal sites, the soft-tissue contrast will be high making it possible to improve contouring accuracy and reduce margins. The potential of the MR-linac lowering treatment toxicity can greatly impact survivorship and quality of life. This would particularly be beneficial for patients diagnosed with cancer in the pelvic region, like prostate cancer, having considerably high chances of survival.

The standard for toxicity monitoring in cancer clinical trials is the prospective clinician reporting of the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE). CTCAE grading, as well as patient-reported outcomes (PRO), is also part of the proposed standard assessment methodology for clinical evaluation of radiotherapy innovations like online MRgRT. Several studies have identified discrepancies between clinician and patient reporting within systemic treatment where clinicians appear to underreport the severity of treatment toxicity, compared to patient-reported severity. Therefore, patient self-reports are an important supplement to the evaluation of online MRgRT as in other oncological settings where they have been used as direct indicators of worsening, persistence or improvement of symptoms and general well-being. Furthermore, patient self-reports reduces the risk of unanticipated treatment toxicities being undetected.

Methods:

Study Design:

The study is a prospective single-arm longitudinal observational study including all prostate cancer patients treated with online MR-guided radiotherapy or CT-guided radiotherapy in the study period.

Participants:

Patients with prostate cancer referred for radiotherapy at Odense University Hospital in the time period 15.11.2020 - 01.07.2022 will be eligible for inclusion.

Data collection:

A patient pathway app, My Hospital, will be used for data collection. A PRO item set for patients with prostate cancer has been developed and tested in a pilot study (PRO-CTCAE and EORTC items). The item set will be used weekly during treatment and 4 weeks following to capture expected and unanticipated symptoms of acute treatment toxicity. During follow-up patients wll be asked to report 8, 12 and 24 weeks after radiotherapy completion. Other questionnaires will be used to measure quality of life (EORTC QLQ-C30+EORTC PR25), health-related quality of life (EQ-5D-5L), patient experience with ePRO (Patient Feedback Form) and patient experience with treatment on a 1.5 T Unity MR-linac (Patient Experience Questionnaire).

Data on clinician management of PROs will be drafted from the patient app My Hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with cancer in the prostate
* referred for primary radiotherapy or salvage radiotherapy

Exclusion Criteria:

* Cognitively unable to provide informed consent
* Unable ro read, understand and complete patient-reported surveys in Danish (electronic or paper-based)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients with prostate cancer and therefore only male participants.
Study Population: Patients receiving radiotherapy (RT) with a curative intent for prostate cancer in the Unity MR-linac or standard linear accelerators using cone-beam CT (CBCT) at Odense University Hospital
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
ACUTE TOXICITY | During or up to six months following radiotherapy completion.
  Mean change in acute urinary and bowel toxicity when treated with MR-guided radiotherapy

SECONDARY OUTCOMES:
QUALITY OF LIFE (QoL) change after CT-guided or online MR-guided radiotherapy | QoL and HRQoL will be reported at baseline (before radiotherapy) and 12 weeks after radiotherapy completion.
  Mean change in QoL from baseline to follow-up week 12. Measured with the questionnaires EORTC QLQ-C30 and Euroqol EQ-5D-5L.
EXPERIENCE | Patient experience will be measured one week following radiotherapy completion.
  The patients are to report how weekly ePROs with real-time feedback in their course of radiotherapy impact their involvement, the quality of care and communication with clinicians. Patient satisfaction is measured with questions from the validated Patient Feedback Form on a 4-point likert scale (strongly agree, agree, disagree, strongly disagree).
ACUTE TOXICITY | Symptoms are reported weekly during treatment and in the four weeks following radiotherapy completion. Patient reporting of acute AEs during follow-up at week 8 and 12 after radiotherapy completion.
  A pelvic item set developed and tested in a pilot study is used to capture symptomatic adverse events (AEs). This item set includes PRO-CTCAE items (5-point likert scale, 0 being absence of symptoms) and EORTC items (4-point likert scale, 1 being absence of symptoms). Median number of weeks to first maximum worsening of the adverse events are measured. Persistence of symptoms is measured as being > baseline score until 12 weeks following radiotherapy.
EXPERIENCE | The patients will be asked to report their experience in the last week of radiotherapy.
  Patient experience with online MR-guided radiotherapy will be measured with a questionnaire specifically developed and validated to capture patient experience in a MR-linac (4-point likert scale).The questionnaire will also be tested on patients undergoing CT-guided radiotherapy to descriptively look at the differences in the two cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Pia KK Møller, MPH, Principal Investigator — Research Unit of Oncology, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Pilot study conducted before this prospective longitudinal study — https://open.rsyd.dk/OpenProjects/openProject.jsp?openNo=775&lang=da